CLINICAL TRIAL: NCT02034955
Title: A Feasibility Study of Post-operative Adaptive Radiation Therapy for Localized Prostate Cancer
Brief Title: Prostatectomy Adaptive Radiation Therapy (ART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 12-5318-C
Record Dates: First submitted 2013-07-03; First posted 2014-01-14 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Adaptive Radiotherapy; Prostatectomy; Patients who had a prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-Operative adaptive radiotherapy (Experimental): All Patients enrolled in this study will have additional scans (Cone-Beam CT, MRI) daily during their treatment. This extra imaging will help us see any changes that might have occurred during radiation treatment and update the treatment plan to include these changes before patient treatment is continued.
  Interventions: Radiation: Post-operative Adaptive Radiation Therapy

INTERVENTIONS:
Radiation: Post-operative Adaptive Radiation Therapy
  Other Names: All Patients enrolled in this study will have additional scans (Cone-Beam CT,MRI) daily during their treatment. This extra imaging will help us see any; changes that might have occurred during radiation treatment and update the treatment plan to include these changes before patient treatment is continued.

SUMMARY:
This study will ultimately aim to evaluate the side effects of treatment by asking 20 subjects to receive post-operative radiotherapy for prostate cancer with the treatment plan adapted after the first week of treatment to account for changes in the target shape. These patients will be asked to complete toxicity scores and a quality of life questionnaire at the start and completion of treatment, and at 3 months 1, 2 and 5 years from the start of radiotherapy. These results will be used to determine the feasibility of the proposed approach, and obtain early estimates of improvements in uncertainty margin requirements for this population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate after radical prostatectomy AND
* Clinical stage pT3, pT4, or pT2 with positive margin OR
* Any p-Stage with a persistently elevated post-operative PSA > 0.05 ng/ml OR
* A delayed rise in PSA post-operatively

Exclusion Criteria:

* Inflammatory bowel disease or other contraindications to radiotherapy
* Prior pelvic radiotherapy
* Previous cytotoxic chemotherapy
* Radiological or pathologic evidence of nodal metastases.
* Planned radiotherapy to pelvic lymph nodes
* Evidence of systemic metastases on imaging.
* Prosthetic hip replacement
* No signed informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change in radiation dose delivered to target volumes and normal tissue | 5 years

SECONDARY OUTCOMES:
Time for radiotherapy replanning | 5 years
Volumetric modulated arc therapy impact in a clinical adaptive Radiotherapy workflow. | 5 years
  Feasibility will be assessed by the time required to perform the adaptive intervention
Toxicity associated with the adaptive radiotherapy technique. | 5 years
  Assessments of gastrointestinal and genitourinary complications using the Common Toxicity Criteria for Adverse Events scoring system and the Expanded Prostate Cancer Index Composite questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Catton, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada